CLINICAL TRIAL: NCT03901703
Title: The Effects of Progressive Functional Ankle Strengthening in Children With Unilateral and Bilateral Spastic Cerebral Palsy
Brief Title: The Effects of Functional Strengthening in Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melek Volkan Yazici (Other)
Responsible Party: Sponsor-Investigator, Melek Volkan Yazici, Principle Investigator, Gazi University
Organization: Gazi University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 465426
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Spastic Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Physical Therapy Modalities; Rehabilitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dorsiflexor Muscle Strengthening Group (Active Comparator): The children in this group will receive functional exercises aiming to strengthen their dorsiflexor muscles alongside standard functional progressive strengthening exercises.
  Interventions: Other: Physiotherapy and Rehabilitation
- Plantarflexor Muscle Strengthening Group (Active Comparator): The children in this group will receive functional exercises aiming to strengthen their plantarflexor muscles alongside standard functional progressive strengthening exercises.
  Interventions: Other: Physiotherapy and Rehabilitation
- Dorsiflexor and Plantarflexor Muscle strengthening Group (Active Comparator): The children in this group will receive functional exercises aiming to strengthen both their dorsiflexor and plantarflexor muscles alongside standard functional progressive strengthening exercises.
  Interventions: Other: Physiotherapy and Rehabilitation

INTERVENTIONS:
Other: Physiotherapy and Rehabilitation — The children in each group will receive 6 weeks of functional strengthening exercises targeting each muscle group according to the arm they are included in.

SUMMARY:
Functional strengthening exercises have been proven to be effective in patients with spastic cerebral palsy. However, which exercise is the most effective is unknown. The aim of this study is to examine the effectiveness of three different progressive functional exercise programs in children with unilateral and bilateral spastic cerebral palsy.

DETAILED DESCRIPTION:
Children with Cerebral Palsy have weakness in thier muscles due to cortical lesions leading to deficiencies in motor control, balance and functional abilities. All children with Cerebral Palsy have shown to present with foot and ankle disorders; the ankle dorsi and plantar flexor muscles are both problematic; the plantarflexors are usually spastic and the dorsiflexors are usually not active enough and usually these muscle problems lead to problems in the childrens' gait abilities. When rehabilitation programs are examined, the results of exercises addressing these problems do not have precise answers. Functional strengthening exercises have been proven to be effective in patients with spastic cerebral palsy. However, which exercise is the most effective is unknown. Which muscle goup has the most effect on gait, balance and functional activities is still unclear. Therefore, the investigator's aim in planning this study is to examine the effectiveness of three progressive functional exercise programs in children with unilateral and bilateral spastic cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Accepting to participate in the study,
* Being between 5-15 years old,
* Having a diagnosis of Spastic Cerebral Palsy,
* Being level I-II according to GMFCS,

Exclusion Criteria:

* Having limited cooperation which prevents participation in the study,
* Refusing to participate in the study,
* Having an orthopedic disorder or systemic illness which prevents movement in the lower extremities,
* Having a Botulinum toxin application in the last 3 months

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2019-01-12 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Pediatric Balance scale | Change of The Pediatric balance scale at 6 weeks.
  The Pediatric Balance Scale is a modified version of the Berg Balance Scale that is used to assess functional balance skills in children. The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points.
Surface Electromyography (sEMG) | Change of sEMG data at 6 weeks.
  Surface electromyography is a non-invasive procedure involving the detection, recording and interpretation of the electric activity of groups of muscles during activity. The procedure is performed using electrodes placed on the skin surface over the muscles to be tested. sEMG is also used to assess the effects of rehabilitation programs and evaluate muscular function in children with cerebral palsy. Due to its non-invasive properties it is safely and widely used in the pediatric population.
The Six minute walk test | Change of 6 MWT at 6 weeks.
  The 6-min walk test (6 MWT) is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes. The 6-minute walk distance (6 MWD) provides a measure for integrated global response of multiple cardiopulmonary and musculoskeletal systems involved in exercise. The test has been shown to be valid and reliable in children with Cerebral Palsy.

CONTACTS AND LOCATIONS:
Overall Officials: Bulent Elbasan, Assoc. Prof., Study Director — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The exercise protocols and results will be shared with other investigators.